CLINICAL TRIAL: NCT06084013
Title: Assessing the Role of Intraoperative Indocyanine Green Perfusion of the Transected Pancreas in Predicting Postoperative Pancreatic Leaks
Brief Title: Use Of Indocyanine Green In Pancreas Surgery
Status: Recruiting | Type: Observational
Sponsor: OHSU Knight Cancer Institute (Other)
Responsible Party: Principal Investigator, Patrick J. Worth, M.D., F.A.C.S., F.S.S.O., Principal Investigator, OHSU Knight Cancer Institute
Other Study IDs: STUDY00025055; NCI-2023-07105 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00025055 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2023-10-02; First posted 2023-10-16 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Carcinoma
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Patients receive indocyanine green IV during surgery, undergo imaging and have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study evaluates the use of indocyanine green to predict postoperative pancreatic leaks in patients undergoing transection of the pancreas.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if altered measurement results of ICG after pancreatectomy is associated with leak rates.

OUTLINE: This is an observational study.

Patients receive indocyanine green intravenously (IV) during surgery, undergo imaging and have their medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* Participant scheduled for open pancreaticoduodenectomy or distal pancreatectomy for any diagnosis
* Participant ≥ 18 years of age
* Ability to understand nature and individual consequences of clinical trial
* Written informed consent from participant or legally authorized representative
* For participants of childbearing potential, a negative pregnancy test and adequate contraception until 14 days after trial intervention
* Participant needs to have an operative drain (any closed suction drain) after the procedure
* Participants that do not require arterial reconstruction
* Participants that require minor portal venous recounstructions including patch venoplasty

Exclusion Criteria:

* Patients with previous history of adverse reaction to contrast dye, ICG or components of the dye
* Prior pancreatectomy
* Known diagnosis of hepatic insufficiency, hepatitis, liver fibrosis or cirrhosis, or chronic pancreatitis
* Because this study focuses on hypoperfusion, patients will be excluded if in postoperative day 3-5 had any of the following: persistent SBP <90 mmHg unresponsive to 1L crystalloid, unexpected ICU transfer, blood transfusion of >2 units intraoperatively or 1 postoperatively, vasopressor treatment or ACLS protocol initiation
* Organ failure, anuria or NSQIP-identified complication will be reviewed by PI and attending surgeon and excluded
* Patients that require arterial reconstruction as part of their procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participant scheduled for open pancreaticoduodenectomy or distal pancreatectomy for any diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of biochemical leak or fistula after pancreatectomy. | Up to 30 days after surgery
  Measurement of drain fluid amylase in post operative period. Defined by definitions of the International Study Group on Pancreatic Surgery (ISGPS) criteria
Perfusion status | During surgical intervention (hours)
  Measured by Indocyanine green (ICG) metrics.

SECONDARY OUTCOMES:
Leak grade via ISGPS classification | Up to 30 days after surgery
  Can be either bile leak, Grade B postoperative pancreatic fistula or grade C postoperative pancreatic fistula
Leak grade by ICG metrics | Up to 30 days after surgery
  ISGPS classification of leak or fistula and the perfusion metrics measures by ICG.
Best practice usage of ICG for pancreatic surgery | Assessed at surgery number 15, approximate 6 months
  Measures through verbal survey to surgeons or OR members

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J Worth, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

REFERENCES:
- [Derived] Salgado-Garza G, Willy A, Rocha FG, Mayo SC, Sheppard BC, Worth PJ. The VIPR-1 trial (Visualizing Ischemia in the Pancreatic Remnant): Assessing the role of intraoperative indocyanine green perfusion in predicting postoperative pancreatic leaks and fistulas: Protocol for a phase II clinical trial. PLoS One. 2025 Jun 24;20(6):e0311025. doi: 10.1371/journal.pone.0311025. eCollection 2025. PMID 40554527